CLINICAL TRIAL: NCT06121752
Title: Device Assisted Full Thickness Resection Versus Endoscopic Submucosal Dissection for Duodenal Neuroendocrine Tumors
Acronym: DNET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, STUDY DIRECTOR, Asian Institute of Gastroenterology, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFTR1
Record Dates: First submitted 2023-10-10; First posted 2023-11-08 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-11

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Device assisted endoscopic full thickness resection (EFTR) (Experimental): The steps of EFTR are as follows. Initially, the lesion will be marked circumferentially using the FTRD probe available with the device (Forced Coag, E1, 20W). Subsequently, wire guided balloon dilatation of the pyloric channel will be performed. The device will be mounted over a therapeutic channel gastroscope and negotiated across the cricopharynx over the guidewire with or without assistance of dilating balloon available with the device. After reaching the target site, the lesion will be pulled withing the FTRD cap with the help of grasping forceps and gentle suctioning. The clip will be fired after ensuring the entry of the lesion inside the cap, the premounted snare closed and electrocautery activated to cut the grasped tissue (HighCut 200W, Effect 4).
  Interventions: Device: EFTR
- Endoscopic submucosal dissection (ESD) (Active Comparator): ESD will be performed using the standard technique under general anaesthesia. The steps of the procedure are as follows: a) marking of the lesion using closed tip of DualKnife J in soft coagulation mode (Effect 4, 80W), b) submucosal lifting injection using saline mixed with indigocarmine dye, c) circumferential mucosal incision (Dry Cut, Effect 2, 30W), d) submucosal dissection (SwiftCoag, Effect 2, 30W), removal of the lesion using suction or a polypectomy snare, f) closure of the defect using endoclips or loop and endoclips.
  Interventions: Procedure: Endoscopic submucosal dissection

INTERVENTIONS:
Procedure: Endoscopic submucosal dissection — Endoscopic resection is recommended for the management of small DNETs measuring ≤10 mm. Various endoscopic techniques have been utilized for the resection of DNETs including endoscopic mucosal resection (EMR), band ligation assisted EMR, endoscopic submucosal dissection (ESD). However, the published studies report a high rate of histologically incomplete resection even with ESD. More recently, device assisted endoscopic full thickness resection (EFTR) has emerged as a safe and effective resection modality in cases with upper and lower gastrointestinal (GI) mucosal as well as submucosal lesions. There is limited data on the outcomes of EFTR in cases with DNETs.
  Arms: Endoscopic submucosal dissection (ESD)
Device: EFTR — Initially, the lesion will be marked circumferentially using the FTRD probe available with the device (Forced Coag, E1, 20W). Subsequently, wire guided balloon dilatation of the pyloric channel will be performed.
  The device will be mounted over a therapeutic channel gastroscope and negotiated across the cricopharynx over the guidewire with or without assistance of dilating balloon available with the device.
  After reaching the target site, the lesion will be pulled withing the FTRD cap with the help of grasping forceps and gentle suctioning.
  The clip will be fired after ensuring the entry of the lesion inside the cap, the premounted snare closed and electrocautery activated to cut the grasped tissue (HighCut 200W, Effect 4).
  Arms: Device assisted endoscopic full thickness resection (EFTR)

SUMMARY:
Introduction :

The incidence of duodenal neuroendocrine tumors (DNETs) is increasing. Endoscopic resection is recommended for the management of small DNETs measuring ≤10 mm. Various endoscopic techniques have been utilized for the resection of DNETs including endoscopic mucosal resection (EMR), band ligation assisted EMR, endoscopic submucosal dissection (ESD). However, the published studies report a high rate of histologically incomplete resection even with ESD. More recently, device assisted endoscopic full thickness resection (EFTR) has emerged as a safe and effective resection modality in cases with upper and lower gastrointestinal (GI) mucosal as well as submucosal lesions. There is limited data on the outcomes of EFTR in cases with DNETs.

In this study, we aim to compare the rate of histologically complete resection (R0) with ESD and EFTR in cases with DNETs.

DETAILED DESCRIPTION:
Primary objective:

Rate of R0 resection in both the groups

Secondary outcomes:

1. Technical success: defined as en-bloc resection of the lesion without any residual lesion endoscopically
2. Procedure duration
3. Adverse Events

Inclusion criteria:

1. Adult patients (≥18 years) with biopsy proven duodenal neuroendocrine tumors (DNETs)
2. Size of the lesion <15 mm
3. Absence of local and distant metastases (EUS and DOTANOC scan)
4. Willing to provide informed consent

Exclusion criteria:

1. Large lesions >15 mm
2. Invasion of muscularis layer and beyond on imaging (EUS)
3. Scarring or deformity in duodenum
4. Active duodenal ulcer
5. History of prior resection
6. Coagulopathy

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years) with biopsy proven duodenal neuroendocrine tumors (DNETs)
2. Size of the lesion <15 mm
3. Absence of local and distant metastases (EUS and DOTANOC scan)
4. Willing to provide informed consent

Exclusion Criteria:

1. Large lesions >15 mm
2. Invasion of muscularis layer and beyond on imaging (EUS)
3. Scarring or deformity in duodenum
4. Active duodenal ulcer
5. History of prior resection
6. Coagulopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Rate of R0 resection in both the groups | 7 days
  Endoscopically and pathologically complete resection

SECONDARY OUTCOMES:
Technical success: defined as en-bloc resection of the lesion without any residual lesion endoscopically | 7 days
  Endoscopically complete resection
Procedure duration | 7 days
  Time to complete each procedure in minutes
Adverse Events | 7 days
  Adverse events during and after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Zaheer Dr Nabi, MBBS MD, Principal Investigator — Asian Institute of Gastroenterology
Locations (1):
- Asian institute of Gastroenterology, Hyderabad, Telangana, India